CLINICAL TRIAL: NCT00681356
Title: A Phase 3, Multicenter, Randomized, Placebo-Controlled, Parallel-Group, Double-Blind Study to Evaluate the Efficacy, Tolerability, Safety, and Pharmacokinetics of 4975 in Patients Undergoing Primary Unilateral Total Knee Arthroplasty
Brief Title: Safety and Efficacy Study of 4975 in Patients Undergoing Total Knee Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anesiva, Inc. (Industry)
Responsible Party: Lisa Renick, CRA, Anesiva, Inc,
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 114-01P
Record Dates: First submitted 2008-05-16; First posted 2008-05-21 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Total Knee Arthroplasty (Replacement)
Keywords: TKA; Total knee arthroplasty; Total knee replacement; Knee surgery
MeSH Terms: interventions — ALGRX-4975

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 4975 - 15 mg
  Interventions: Drug: 4975, 15 and 5 mg
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Comparator
- 3 (Experimental): 4975 - truncated for Phase 3
  Interventions: Drug: 4975 - 5 mg

INTERVENTIONS:
Drug: 4975, 15 and 5 mg — Direct instillation into the surgical site
  Other Names: Adlea
  Arms: 1
Drug: Placebo Comparator — Direct instillation into the surgical site
  Arms: 2
Drug: 4975 - 5 mg — Direct instillation into the surgical site
  Arms: 3

SUMMARY:
Evaluate the efficacy, tolerability, safety, and pharmacokinetics of 4975 in patients undergoing total knee replacement

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy, tolerability, safety, and pharmacokinetics of 4975 in patients undergoing primary unilateral total knee arthroplasty

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged 18 to 85 years with an American Society of Anesthesiologists (ASA) status of I, II, or III
* Planning to undergo primary unilateral Total Knee Arthroplasty (TKA)

Key Exclusion Criteria:

* A body mass index (BMI) greater than 43
* Known bleeding disorder or is taking agents affecting coagulation preoperatively
* Use of medications or a medical condition that in the investigator's opinion could adversely impact the patient's participation or safety, conduct of the study, or interfere with the pain assessments
* Diabetes mellitus with a known HbA1C>9.5 or a history of prolonged uncontrolled diabetes
* Previous knee arthroplasty (partial or total) of the same knee
* Participated in another clinical trial within 30 days prior to the planned TKA surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) measures of pain at prespecified times | Primary endpoint is 2 days (4-48 hours)

SECONDARY OUTCOMES:
Other efficacy parameters, safety and tolerability of 4975 | 42 Days or Early Termination

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Comfort, MD, Study Director — Anesiva, Inc.
Locations (25):
- United States (25):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Springhill Medical Center, Mobile, Alabama
  - Hellen Keller Hospital, Sheffield, Alabama
  - Visions Clinical Research/Tucson Medical Center, Tucson, Arizona
  - Glendale Adventist Medical Center - Lotus Clinical Research, Glendale, California
  - Physicians Clinical Research Corporation, Laguna Hills, California
  - Saddleback Memorial Medical Center/Accurate Clinical Trials, Laguna Hills, California
  - Webster Orthopeadic Medical Group, Oakland, California
  - UCSF-Mt. Zion Medical Center, San Francisco, California
  - Orthopedic Associates of Hartford, Hartford, Connecticut
  - Florida Hospital - Florida Research Associates, LLC, DeLand, Florida
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Miami Institute for Medical Research, Miami, Florida
  - Southeastern Clinical Research Consultants, Orlando, Florida
  - Coastal Medical Research, Port Orange, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Ruxton Professional Center - Orthopaedic Associates, Towson, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Sewickley Valley Hospital, Sewickley, Pennsylvania
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Memorial City Hospital - Memorial Hermann Healthcare System, Houston, Texas

REFERENCES:
- [Derived] Hartrick CT, Pestano C, Carlson N, Hartrick S. Capsaicin instillation for postoperative pain following total knee arthroplasty: a preliminary report of a randomized, double-blind, parallel-group, placebo-controlled, multicentre trial. Clin Drug Investig. 2011 Dec 1;31(12):877-82. doi: 10.1007/BF03256925. PMID 21971213
- See also: Anesiva, Inc. Home Page — http://www.anesiva.com/wt/page/pipeline
- See also: ADLEA Product Information — http://www.anesiva.com/wt/page/adlea